CLINICAL TRIAL: NCT04545801
Title: Ketamine for Analgesia After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor, head of department of anesthesia and critical care, Mongi Slim Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ketamine cesarean
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Cesarean Section; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine Group (Active Comparator): Patients recieving 0.25 mg/kg of ketamine 5 minutes after spinal anesthesia
  Interventions: Drug: 0.25 mg/kg of Ketamine
- Placebo Group (Placebo Comparator)
  Interventions: Drug: 20ml of normal saline solution

INTERVENTIONS:
Drug: 0.25 mg/kg of Ketamine — patients will recieve 0.25mg/kg of ketamine intravenously 5 min after spinal anesthesia
  Arms: Ketamine Group
Drug: 20ml of normal saline solution — 20ml of normal saline solution intravenously 5 minutes after spinal anesthesia
  Arms: Placebo Group

SUMMARY:
In this prospective randomized trial, investigators compared the analgesic effect of subanesthetic dose of ketamine versus placebo in parturients undergoing cesarean section under spinal anesthesia.

DETAILED DESCRIPTION:
In this prospective randomized trial, investigators compared the analgesic effect of subanesthetic dose of ketamine versus placebo in parturients undergoing cesarean section under spinal anesthesia.

The patients were randomized in two groups:

* Group Ketamine: these patients recieved 0.25 mg/kg of Ketamin intravenously 5 minutes after the spinal anesthesia.
* Group Placebo: recieved 20 ml of normal saline solution intravenously 5 minutes after the spinal puncture.

The investigators recorded intra demographic, intraoperative and post operative data.

The main outcome was the analgesic score: the visual analog scale (VAS). dynamic VAS was also monitored at 24 hours post operatively.

ELIGIBILITY:
Inclusion Criteria:

* full term pregnant adult patients
* Monofetal pregnancy
* scheduled for urgent or elective cesarean section under spinal anesthesia

Exclusion Criteria:

* necessity of general anesthesia during the procedure
* Post partum hemorrage

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — including only female patients undergoing cesarean section
Enrollment: 80 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Dynamic Visual Analog Scale | 24 hours after cesarean section
  Pain score VAS range from 0 to 10, high scores mean worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Mongi Slim University Hospital, La Marsa, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No